CLINICAL TRIAL: NCT05331937
Title: Transcranial Magnetic Stimulation (TMS) for Patients With Exposure Therapy-resistant Obsessive-compulsive Disorder (OCD): TETRO - a Multicenter Randomized Controlled Trial
Brief Title: TMS for Exposure Therapy Resistant OCD
Acronym: TETRO
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: GGZ inGeest (Other); Radboud University Medical Center (Other); ProPersona (Other); Maastricht University Medical Center (Other); Mondriaan (Unknown); Neurocare (Other)
Responsible Party: Principal Investigator, O.A. van den Heuvel, prof.dr. (MD PhD), Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021.0670 - NL78930.029.21
Record Dates: First submitted 2022-03-29; First posted 2022-04-18 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: 1 Hz Real rTMS to the Pre-SMA; 1 Hz Sham rTMS to the Pre-SMA
MeSH Terms: interventions — Transcranial Magnetic Stimulation; Implosive Therapy

STUDY DESIGN:
Intervention Model Description: multi-center placebo-controlled double-blind randomized controlled trial with an intervention phase of 5-7 weeks and a follow-up phase of 12 months
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- real rTMS (Experimental): verum rTMS condition, 1500 continuous 1-Hz pulses to the pre-SMA
  Interventions: Combination Product: repetitive transcranial magnetic stimulation (rTMS)
- sham rTMS (Sham Comparator): sham rTMS condition, 1500 continuous 1-Hz pulses to the pre-SMA
  Interventions: Combination Product: repetitive transcranial magnetic stimulation (rTMS)

INTERVENTIONS:
Combination Product: repetitive transcranial magnetic stimulation (rTMS) — rTMS (real versus sham) is used as adjuvant to ERP
  Other Names: exposure therapy with response prevention (ERP)

SUMMARY:
TETRO is a multi-center placebo-controlled double-blind randomized controlled trial with an intervention phase of 5-7 weeks and a follow-up phase of 12 months in 250 adult (18 years and older) OCD patients who show no/insufficient response to ERP, aiming to establish the cost-effectiveness of low frequency (1 Hz) rTMS to the pre-SMA (compared to sham rTMS to the pre-SMA) as adjuvant treatment to exposure with response prevention (ERP). The treatment consists of 4 times/week rTMS combined with ERP for at least 5 weeks (20 sessions), with optional extension phase of 1 or 2 weeks (maximum of 28 sessions in total).

DETAILED DESCRIPTION:
Rationale:

Obsessive-compulsive disorder (OCD) is a serious and disabling mental disorder, characterized by obsessions and compulsions and associated with substantial comorbidity and morbidity (Stein et al. 2019). Approximately 50% of patients treated with standard treatments (exposure therapy with response prevention (ERP) with/without medication) fail to respond fully, resulting in chronicity and poor participation in social and educational/occupational domains. We propose to fill the gap between the standard treatments (exposure therapy with/without medication) on the one side and invasive end-stage strategies (brain surgery) on the other side, using a non-invasive alternative: repetitive transcranial magnetic stimulation (rTMS). Despite proven efficacy (Zhou et al. 2017; Rehn et al. 2018; Fitzsimmons et al. 2022), rTMS for OCD is not yet covered by the Dutch insurance system while rTMS for treatment resistant depression is. This multi-center randomized controlled trial, supported by the 'veelbelovende zorg' grant of Zorg Instituut Nederland (ZIN), aims to establish the added value of rTMS applied over the pre-supplementary motor area (preSMA) when combined with ERP in OCD patients, who show no/insufficient response to ERP (alone or combined with medication). In case of proven cost-effectiveness it will lead to the addition of rTMS as insured health care for patients with OCD.

Objective: assess the (cost-)effectiveness of 1Hz rTMS to the pre-SMA as adjuvant treatment to ERP in OCD patients who show no/insufficient response to ERP (alone or combined with medication)

Study design: multi-center placebo-controlled double-blind randomized controlled trial with an intervention phase of 5-7 weeks and a follow-up phase of 12 months

Study population: 250 adult (18 years and older) OCD patients who show no/insufficient response to ERP

Intervention (if applicable): Low frequency (1 Hz) rTMS to the pre-SMA (compared to sham rTMS to the pre-SMA) as adjuvant treatment to ERP, 4 times/week for at least 5 weeks (20 sessions), with optional extension phase of 1 or 2 weeks (maximum of 28 sessions in total)

Main study parameters/endpoints: the pre-versus-post-treatment standardized mean difference (SMD) in severity of OCD (Yale-Brown Obsessive-Compulsive Scale - Y-BOCS), version 2. The post-treatment Y-BOCS score will be obtained at the end of treatment, i.e, after 20, 24 or 28 sessions.

Secondary study parameters/endpoints:

* Response (≥35% reduction on Y-BOCS-v2) and remission (Y-BOCS≤12) as established through international expert opinion
* Standard Mean Difference (SMD) on the Clinical Global Impression (CGI) severity scale
* Clinical Global Impression (CGI) improvement scale
* Quality of life (EQ-5D-5L)
* Societal costs, measured through the iMTA Productivity Cost Questionnaire (iPCQ) and the iMTA Medical Consumption Questionnaire (iMCQ)
* Depression, measured using the Beck Depression Inventory (BDI) at baseline, post-treatment and follow-up. In addition we will administer a visual analogue scale (VAS) for depression at these same time points, plus every week during treatment, to monitor the effects of treatment on severity of depressive symptoms.
* Anxiety, measured using the Beck Anxiety Inventory (BAI) and a VAS; following the same procedure and rationale as for depression.
* Tolerability of the treatment and side effects, using an in-house questionnaire

Exploratory outcomes and/or influencing factors:

* Patient adherence to treatment protocol, as measured using the Patient Exposure and Response Prevention Adherence Scale (PEAS)
* Difference between responders and non-responders on circadian rhythm and sleep disorders at baseline as defined by the Holland Sleep Disorders Questionnaire (HSDQ).
* Structural brain network characteristics (using T1 and diffusion weighted scans) to predict treatment response / relapse.
* Functional resting-state and task-based (during emotional processing) brain network characteristics (using echo-planar imaging) to predict treatment response / relapse.
* Variation in the exact stimulation location as ascertained and recorded by neuronavigation in relation to treatment outcome.
* Contribution of demographic and clinical variables (sex, age, medication status) and pre-existing comorbidities (i.e. comorbid tics, depression, anxiety, autism) to the variance in treatment outcome.
* In OCD patients with comorbid tics: tic severity, measured using the Yale Global Tic Severity Scale (Y-GTSS).
* Variation in treatment expectancy (7-items credibility and expectancy questionnaire (CEQ)) and blinding success (1-item question 'in which condition do you think you were?') in relation to treatment outcome.

ELIGIBILITY:
Inclusion Criteria:

* OCD as current primary diagnosis
* Age 18 and older
* Yale-Brown Obsessive-Compulsive Scale (YBOCS) score of 16 or higher.
* Insufficient response to state-of-the art exposure therapy with response prevention (ERP) and/or drop-out from ERP due to extreme anxiety/avoidance
* The following comorbid disorders are allowed (as long as OCD is the current primary diagnosis): depression, other anxiety disorders, ADHD, tic/Tourette's disorder, eating disorders, personality disorders, autism spectrum disorder (when this does not dominate the clinical profile, i.e. is not main diagnosis).
* Commitment to actively undergo intensive exposure therapy (both supervised during ERP sessions, as well as unsupervised at home)
* Unmedicated (for at least 8 weeks) or stable dosage of psychotropic medication (for at least 8 weeks), involving serotonergic antidepressants (SSRI, SNRI, clomipramine). Other psychotropic medication that is allowed (provided dosage is stably established for at least 8 weeks): methylphenidate, mood stabilizers, antipsychotic drugs
* Ability to participate in frequent treatment sessions (4 days/week, for 5 (or 6, or 7) weeks) at one of the 5 sites nearest to their home and/or work
* Ability to participate in pre-treatment MRI session (for neuronavigation) at one of the 3 academic sites nearest to their home and/or work
* Capacity for providing informed consent

Exclusion Criteria:

* OCD patients with hoarding as main symptom dimension
* The following comorbid disorders (current diagnosis) are not allowed: psychotic disorders, bipolar disorder, autism spectrum disorder (when this dominates the clinical profile, i.e. is diagnosed as main disorder), substance use disorder
* Active suicidal thoughts and intent to act on it
* Chronic use of benzodiazepines is not allowed
* Cochlear implant
* (History of) epilepsy
* Pregnancy
* Extreme claustrophobia or metallic objects in or on the body, preventing from participation in MRI session
* Space-occupying lesion on MRI
* Previous rTMS treatment (for blinding reasons)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2022-05-16 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
YBOCS-2 | baseline (T0) versus directly post-treatment (5, 6 or 7 weeks post-baseline, dependent on duration of treatment)
  pre-versus-post-treatment standardized mean difference (SMD) in severity of OCD as measured with the Yale-Brown Obsessive-Compulsive Scale (version 2)

SECONDARY OUTCOMES:
response and remission | baseline (T0) versus directly post-treatment (5, 6 or 7 weeks post-baseline, dependent on duration of treatment) + 3, 6 and 12 months follow-up
  response: ≥35% reduction on Y-BOCS | remission: Y-BOCS≤12
Standard Mean Difference (SMD) on the Clinical Global Impression (CGI) severity scale | baseline (T0) versus directly post-treatment (5, 6 or 7 weeks post-baseline, dependent on duration of treatment) + 3, 6 and 12 months follow-up
  global functioning
Clinical Global Impression (CGI) improvement scale | baseline (T0) versus directly post-treatment (5, 6 or 7 weeks post-baseline, dependent on duration of treatment) + 3, 6 and 12 months follow-up
  global improvement
Quality of life (EQ-5D-5L) | baseline (T0) versus directly post-treatment (5, 6 or 7 weeks post-baseline, dependent on duration of treatment) + 3, 6 and 12 months follow-up
  quality of life
Societal costs, measured through the iMTA Productivity Cost Questionnaire (iPCQ) | baseline (T0) versus directly post-treatment (5, 6 or 7 weeks post-baseline, dependent on duration of treatment) + 6 and 12 months follow-up
  cost effectiveness
Societal costs, measured through the iMTA Medical Consumption Questionnaire (iMCQ) | baseline (T0) versus directly post-treatment (5, 6 or 7 weeks post-baseline, dependent on duration of treatment) + 6 and 12 months follow-up
  cost effectiveness
depression, measured through the Beck Depression Inventory | baseline (T0) versus directly post-treatment (5, 6 or 7 weeks post-baseline, dependent on duration of treatment) + 3, 6 and 12 months follow-up
  comorbid depression
anxiety, measured through the Beck Anxiety Inventory | baseline (T0) versus directly post-treatment (5, 6 or 7 weeks post-baseline, dependent on duration of treatment) + 3, 6 and 12 months follow-up
  comorbid anxiety
Tolerability of the treatment and side effects, using an in-house questionnaire | after 1st and last week of treatment
  tolerability and side effects

OTHER OUTCOMES:
tic severity, measured using the Yale Global Tic Severity Scale (YGTSS) | baseline (T0) versus directly post-treatment (5, 6 or 7 weeks post-baseline, dependent on duration of treatment) + 3, 6 and 12 months follow-up
  tic severity (only in OCD patients with comorbid tics)

CONTACTS AND LOCATIONS:
Locations (8):
- Netherlands (8):
  - Amsterdam UMC, location VU Medical Center, Amsterdam, North Holland
  - GGZ inGeest, Amsterdam
  - Neurocare, Eindhoven
  - Neurocare, Groningen
  - Maastricht UMC+, Maastricht
  - Mondriaan, Maastricht
  - ProPersona, Nijmegen
  - Radboudumc, Nijmegen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fitzsimmons SMDD, van der Werf YD, van Campen AD, Arns M, Sack AT, Hoogendoorn AW; other members of the TETRO Consortium; van den Heuvel OA. Repetitive transcranial magnetic stimulation for obsessive-compulsive disorder: A systematic review and pairwise/network meta-analysis. J Affect Disord. 2022 Apr 1;302:302-312. doi: 10.1016/j.jad.2022.01.048. Epub 2022 Jan 15. PMID 35041869
- [Background] Rehn S, Eslick GD, Brakoulias V. A Meta-Analysis of the Effectiveness of Different Cortical Targets Used in Repetitive Transcranial Magnetic Stimulation (rTMS) for the Treatment of Obsessive-Compulsive Disorder (OCD). Psychiatr Q. 2018 Sep;89(3):645-665. doi: 10.1007/s11126-018-9566-7. PMID 29423665
- [Background] Zhou DD, Wang W, Wang GM, Li DQ, Kuang L. An updated meta-analysis: Short-term therapeutic effects of repeated transcranial magnetic stimulation in treating obsessive-compulsive disorder. J Affect Disord. 2017 Jun;215:187-196. doi: 10.1016/j.jad.2017.03.033. Epub 2017 Mar 18. PMID 28340445
- [Background] Stein DJ, Costa DLC, Lochner C, Miguel EC, Reddy YCJ, Shavitt RG, van den Heuvel OA, Simpson HB. Obsessive-compulsive disorder. Nat Rev Dis Primers. 2019 Aug 1;5(1):52. doi: 10.1038/s41572-019-0102-3. PMID 31371720